CLINICAL TRIAL: NCT06197958
Title: Comparison of Concentric-eccentric Exercises in Patellofemoral Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0455
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Patello Femoral Syndrome; Patellofemoral Pain; Knee Pain Chronic
Keywords: concentric excercise; eccentric excercise; Iliotibial Band
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Intervention Model Description: randomized clinical trail
Who Masked: Outcomes Assessor
Masking Description: the assessor who will take the readings is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eccentric exercises (Experimental): Group A: Group A will receive 3 sets of eccentric exercises with 10 RM (repetition maximum) in six sessions.
  Interventions: Other: eccentric exercises
- concentric exercises (Experimental): Group B: Group B will receive 3 sets of concentric exercises with 10 RM in six sessions
  Interventions: Other: concentric exercises

INTERVENTIONS:
Other: eccentric exercises — eccentric exercises like walking down stairs, lowering a weight during shoulder press, the downward motion of squatting, the downward motion of a push-up, lowering the body during a crunch, lowering the body during a pull-up 3 sets with 10 RM (repetition maximum) for six week training.
  Arms: eccentric exercises
Other: concentric exercises — concentric exercises like walking upstairs, pushing up in a bench press, the beginning portion of a deadlift when you lift the barbell off the ground, sitting up in a sit up, pushing up from a lowered push-up and standing up in a back squat 3 sets with 10 RM.
  Arms: concentric exercises

SUMMARY:
Patellofemoral pain syndrome is due to dysfunctional dynamic knee valgus resulting from decrease in strength of hip abductors or abnormal rear-foot eversion with pes pronatus valgus. It is also associated with vastus medialis/vastus lateralis disbalance, hamstring tightness or iliotibial tract tightness.

DETAILED DESCRIPTION:
Patellofemoral pain syndrome is due to dysfunctional dynamic knee valgus resulting from decrease in strength of hip abductors or abnormal rear-foot eversion with pes pronatus valgus. It is also associated with vastus medialis/vastus lateralis disbalance, hamstring tightness or iliotibial tract tightness. The pain is felt around or behind the patella. The causes are multifactorial. A decline in ability to perform physical activity is seen. The aim of this study will be to compare the effects of concentric and eccentric exercises on pain, strength and ROM in patellofemoral pain syndrome.A randomized clinical trial will be performed at Barki Advance Physiotherapy Center Multan through convenience sampling technique on 24 patients which will be allocated through random sampling through sealed opaque enveloped into group A and group B. Group A will receive eccentric exercises like walking down stairs, lowering a weight during shoulder press, the downward motion of squatting, the downward motion of a push-up, lowering the body during a crunch, lowering the body during a pull-up 3 sets with 10 RM (repetition maximum) for six week training. The group B will receive concentric exercises like walking upstairs, pushing up in a bench press, the beginning portion of a deadlift when you lift the barbell off the ground, sitting up in a sit up, pushing up from a lowered push-up and standing up in a back squat 3 sets with 10 RM. Screening tools include patellar grind test with positive Clark's sign and VAS (visual analogue scale) for pain rating. Outcomes will be measured through knee resisted test and MMT grading for knee extensor/flexor strength and goniometer for ROM. Data will be analyzed using SPSS software version 25. After assessing normality, it will be decided either parametric or non parametric test will be used within a group or between two groups. Effectiveness of concentric and eccentric exercises will be analyzed by comparison in individuals with patellofemoral pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Players between the age 18 to 36 years.
* Both male and female gender.
* Patients who have Patellar grind test positive.
* The presence of retropatellar or peripatellar pain.
* Reproduction of retropatellar or peripatellar pain with squatting, stair climbing, prolonged sitting, or other functional activities loading the PFJ in a flexed position.

Exclusion Criteria:

* Individuals with a history of recent trauma or surgery of lower limb (16), administration of steroid injection in the past 6 months.
* Recent administration of platelet-rich plasma containing growth factors, diagnosis of rheumatoid arthritis, myositis ossificans, diagnosis of other muscular disorder.
* Patients who had taken physical therapy of any sort in the past six months will be excluded from the study.
* Furthermore, individuals with any history of occupation-related pain will be ruled out

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
patellofemoral pain | pre and 6 weeks post interventional
  pain is measured by VAS (Visual Analogue Scale)
range of motion | pre and 6 weeks post interventional
  ROM is measured by goniometer
knee extensor/flexor strength | pre and 6 weeks post interventional
  knee extensor/flexor strength is measured by knee resisted test and MMT grading

CONTACTS AND LOCATIONS:
Overall Officials: moiz kamal, DPT, Principal Investigator — study principal investigator
Locations (1):
- barki advance physiotherapy center Multan, Multan Khurd, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crossley KM, Stefanik JJ, Selfe J, Collins NJ, Davis IS, Powers CM, McConnell J, Vicenzino B, Bazett-Jones DM, Esculier JF, Morrissey D, Callaghan MJ. 2016 Patellofemoral pain consensus statement from the 4th International Patellofemoral Pain Research Retreat, Manchester. Part 1: Terminology, definitions, clinical examination, natural history, patellofemoral osteoarthritis and patient-reported outcome measures. Br J Sports Med. 2016 Jul;50(14):839-43. doi: 10.1136/bjsports-2016-096384. Epub 2016 Jun 24. No abstract available. PMID 27343241
- [Background] Glaviano NR, Kew M, Hart JM, Saliba S. DEMOGRAPHIC AND EPIDEMIOLOGICAL TRENDS IN PATELLOFEMORAL PAIN. Int J Sports Phys Ther. 2015 Jun;10(3):281-90. PMID 26075143
- [Background] Petersen W, Ellermann A, Gosele-Koppenburg A, Best R, Rembitzki IV, Bruggemann GP, Liebau C. Patellofemoral pain syndrome. Knee Surg Sports Traumatol Arthrosc. 2014 Oct;22(10):2264-74. doi: 10.1007/s00167-013-2759-6. Epub 2013 Nov 13. PMID 24221245
- [Result] Smith BE, Selfe J, Thacker D, Hendrick P, Bateman M, Moffatt F, Rathleff MS, Smith TO, Logan P. Incidence and prevalence of patellofemoral pain: A systematic review and meta-analysis. PLoS One. 2018 Jan 11;13(1):e0190892. doi: 10.1371/journal.pone.0190892. eCollection 2018. PMID 29324820